CLINICAL TRIAL: NCT07235111
Title: Omics Sciences for the Identification of Pathogenetic Mechanisms and Biomarkers in Neurodegenerative Diseases
Acronym: NeurOmics
Status: Recruiting | Type: Observational
Sponsor: Ospedale Policlinico San Martino (Other)
Collaborators: Istituto Italiano di Tecnologia (Other)
Responsible Party: Sponsor
Other Study IDs: Neuromics (209/2024 id.:13896)
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-02

CONDITIONS: Alzheimer Disease; FTD; Young-onset Dementia; MCI; Parkinson Disease; ALS (Amyotrophic Lateral Sclerosis)
Keywords: LEWY BODIES DISEASE; young-onset dementia; alzheimer; parkinson; als; mci
MeSH Terms: conditions — Alzheimer Disease; Parkinson Disease; Amyotrophic Lateral Sclerosis; Neurocognitive Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood, saliva, PBMCs (Peripheral blood mononuclear cells), plasma, serum and/or urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with neurodegenerative diseases: The study aims to identify pathogenic genomic variants and/or altered molecular pathways in these patients by analysing the entire genome and integrating these data with gene expression data and/or epigenomic and/or protein expression data. The study also aims to identify new markers for the diagnosis and monitoring of neurodegenerative diseases by analysing collected biological samples such as blood and blood derivatives, including liquid biopsy approaches using the most advanced technologies available at the t

SUMMARY:
The study aims to use 'omics' sciences, employing the most advanced technologies currently available, in order to identify pathogenic genomic variants, proteins and/or altered molecular pathways in neurodegenerative diseases and to obtain a new and more complete characterisation of subjects affected by the neurodegenerative diseases under study. Thanks to the integration of genomic, gene expression (transcriptomic and epigenomic), protein and metabolic data and clinical data, the study also aims to identify new markers for the diagnosis, prognosis, also in terms of response to therapy, and monitoring of neurodegenerative diseases.

The study involves the enrolment of at least 1.200 individuals with neurodegenerative disease.

DETAILED DESCRIPTION:
The study aims to use 'omics' sciences, employing the most advanced technologies currently available, in order to identify pathogenic genomic variants, proteins and/or altered molecular pathways in neurodegenerative diseases and to obtain a new and more complete characterisation of subjects affected by the neurodegenerative diseases under study. Thanks to the integration of genomic, gene expression (transcriptomic and epigenomic), protein and metabolic data and clinical data, the study also aims to identify new markers for the diagnosis, prognosis, also in terms of response to therapy, and monitoring of neurodegenerative diseases.

The study involves the enrolment of at least 1.200 individuals with neurodegenerative disease.

The study population consists of patients with neurodegenerative diseases from the IRCCS Ospedale Policlinico San Martino in Genoa and the IRCCS Cà Granda Ospedale Maggiore Policlinico Foundation in Milan and any other units that may wish to participate in the study after approval by the EC. The subjects eligible for enrolment will be identified during the outpatient visits scheduled during the clinical controls at the two centres. During these visits, patients will be proposed to participate in the study. The clinical diagnosis will be made according to the criteria used for each subtype of neurodegenerative disease and detailed in the project.

Different types of biological samples will be collected from patients enrolled in the study, mainly peripheral blood, saliva (if blood sampling is not possible) and urine. Samples will be taken during regular sampling at one of the follow-up visits.

Omics' analyses, mainly genomics, transcriptomics, epigenomics, etc., will be performed on the biological samples taken and/or their derivatives.

Analyses may be performed on genetic material extracted from whole peripheral blood, saliva, PBMCs (Peripheral blood mononuclear cells), plasma, serum and/or urine.

An aliquot of DNA, pseudonymised, will be sent to the Laboratories of the Italian Institute of Technology (Genoa and Aosta) for genome and other omics analysis.

An aliquot of DNA and the derivatives from the collection (serum, plasma, PBMC) will be stored in the Biobank of the Clinical Centres to which the patients are referred.

The study does not foresee the use of experimental drugs or other interventions on the patient, other than those foreseen in the diagnostic routine.

The study plans to characterise from an 'omics' point of view about 1.200 patients affected by neurodegenerative diseases and afferent to the IRCCS Policlinico San Martino in Genoa and to the Fondazione IRCCS Policlinico Cà Granda in Milan and any other Units that may wish to participate in the study after approval by the relevant TEC.

The aim of the Study, for the different pathologies of interest, is to identify, through the study of the genome, single and polygenic variants, both rare and common, single nucleotide (SNV) and/or structural (such as, CNV, insertions, translocations, inversions and mobile element insertions (MEI)) that may be causative or confer an increased risk of developing the disease. Furthermore. the integration of genomic data with other 'omics' sciences will make it possible to correlate the presence of such variations with gene, protein and metabolic expression, to delineate different trajectories of molecular mechanisms associated with neurodegeneration, their impact on disease progression and the identification of new therapeutic targets.

ELIGIBILITY:
Inclusion Criteria

• Patients suffering from neurodegenerative diseases

Exclusion Criteria

• Patients not suffering from neurodegenerative diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NeurOmics is a multicenter observational study, conducted on patients diagnosed with neurodegenerative disease (AD, MCI, PD, ALS, atypical parkinsonisms)
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2034-09-17 (Estimated); Study Completion 2039-09-17 (Estimated)

PRIMARY OUTCOMES:
Identify variants in our genetic makeup, proteins, and/or altered metabolic pathways in patients with neurodegenerative diseases | 10 years
  Thanks to the integration of genomic, gene expression, protein and metabolic data and clinical data, the Firm aims to identify new markers for diagnosis, prognosis, also in terms of response to therapy, and monitoring of neurodegenerative diseases. There will be three outcomes from the study.
  * Identification of variants in our coding DNA (i.e. that serves to produce proteins needed by our cells) that are known to cause or predispose to Alzheimer's disease;
  * Analyze the non-coding regions of our DNA (i.e. regions that serve to regulate, modify, inhibit the production of proteins in our body) in search of variants that can cause, modify the prognosis and/or response to drugs in Alzheimer's disease;
  * Investigate the role of genetic-molecular alterations on the clinical phenotype for the most frequent variants

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Policlinico San Martino, Genoa, Genoa, Italy

DOCUMENTS (1):
  • Study Protocol (2023-11-30): https://cdn.clinicaltrials.gov/large-docs/11/NCT07235111/Prot_000.pdf